CLINICAL TRIAL: NCT03086408
Title: The Safety and Efficacy of the Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) for Short Diagnostic Bronchoscopy Procedures
Brief Title: Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) and Diagnostic Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vladimir Nekhendzy, Clinical Professor of Anesthesiology and Otolaryngology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 40295
Record Dates: First submitted 2017-03-06; First posted 2017-03-22 (Actual); Results first posted 2020-06-23 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Bronchoscopy
Keywords: airway management; high flow nasal oxygen; high flow nasal cannula; THRIVE
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- THRIVE (Experimental): high flow nasal oxygen
  Interventions: Device: THRIVE
- endotracheal tube or supraglottic airway (Active Comparator): tracheal intubation or supraglottic airway device
  Interventions: Device: Endotracheal tube or Supraglottic airway

INTERVENTIONS:
Device: THRIVE — active nasal oxygen delivery system
  Arms: THRIVE
Device: Endotracheal tube or Supraglottic airway — Plastic devices for mechanical ventilation
  Arms: endotracheal tube or supraglottic airway

SUMMARY:
The purpose of this study is to investigate whether diagnostic bronchoscopy can be safely and potentially more effectively performed without the use of tracheal intubation or a supraglottic airway, under completely unobstructed surgical conditions afforded by THRIVE: Transnasal Humidified Rapid- Insufflation Ventilatory Exchange. THRIVE provides patient's gas exchange through rapid insufflation of high-flow oxygen via specialized nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for diagnostic bronchoscopy

Exclusion Criteria:

* Patients with significantly decreased myocardial function (ejection fraction < 50%)
* Patients with abnormal cardiac rhythm and conduction abnormalities, except for patients with isolated, asymptomatic premature atrial and ventricular contractions.
* Patients with significant peripheral vascular disease, such as those with the symptoms of intermittent claudication.
* Patients with known significant cerebrovascular disease, such as history of cerebrovascular accidents (CVAs) and transient ischemic attacks (TIAs).
* Patients with significant renal insufficiency, as manifested by estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2.
* Patients with electrolyte (K+, Ca++) abnormalities, as determined by the lab values outside of a normal range.
* Patients with the history or symptoms of increased intracranial pressure or reduced intracranial compliance (e.g. headaches, nausea and vomiting, visual changes, mental changes).
* Patients with skull base defects.
* Patients with pulmonary hypertension who have pulmonary artery pressures above the normal range.
* Patients with significant chronic obstructive or restrictive lung diseases, as manifested by known history of baseline chronic hypoxia and/or hypercapnia, and/or baseline room air SpO2 < 95%.
* Obese patients with BMI above 35 kg/m2.
* Patients with severe and poorly controlled gastroesophageal reflux disease despite medical treatment.
* Patients with hiatal hernia and full stomach patients.
* Patients on immunosuppressive medications.
* Patient's refusal to participate in the study.
* Patients who do not understand English or mentally handicapped.
* Pregnant or breastfeeding patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Nekhendzy, MD, Study Chair — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- THRIVE: Participants receive Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) active nasal oxygen delivery system.
- Endotracheal Tube or Supraglottic Airway: Participants receive tracheal intubation or supraglottic airway device for mechanical ventilation.
Period: Overall Study
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- THRIVE: Participants receive THRIVE active nasal oxygen delivery system.
- Total: Total of all reporting groups
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (19.01) | 56.5 (16.17) | 55.0 (17.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Lowest Intraoperative Peripheral Oxygen Saturation (SpO2)
Description: Peripheral oxygen saturation is an estimate of the amount of oxygen in the blood.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: percentage of oxygen
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
percentage of oxygen | 94.7 (6.65) | 98.7 (1.70)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = -4, 95% CI 2-sided [-9.00 to 1.00]

2. Primary Outcome: Awakening/Extubation Time
Description: Recorded from the end of surgery until the return of patient's protective airway reflexes and patient opening eyes to command.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
minutes | 10.1 (2.42) | 9.2 (4.87)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-2.89 to 4.69]

3. Primary Outcome: Time to Bronchoscope Placement in Trachea
Description: Recorded from the moment of the introduction of the bronchoscope in patient's mouth to tracheal placement.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
minutes | 1.03 (0.38) | 1.1 (0.68)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 0.78, t-test, 2 sided; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.61 to 0.47]

4. Primary Outcome: Number of Tracheal Bronchoscope Placements Required
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: placements
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
placements | 0.2 (0.42) | 0.6 (1.07)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 0.30, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.30 to 0.50]

5. Primary Outcome: Duration of Procedure
Description: Recorded from the introduction of the bronchoscope in patient's mouth to withdrawing the bronchoscope at the completion of procedure.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
minutes | 15.6 (7.90) | 15.5 (11.17)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 0.98, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-8.62 to 8.82]

6. Secondary Outcome: Time to Patient Being Alert and Oriented x 4
Description: Recorded from patient's admission to the post-anesthesia care unit (PACU) to patient's orientation to person, place, time, and situation as assessed by the recovery room nurse.
Time Frame: Duration of surgery (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
minutes | 1.2 (3.12) | 0.67 (0.87)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-1.64 to 2.84]

7. Secondary Outcome: Recovery Room Discharge-ready Time
Description: From admission to recovery room, to discharge from recovery room
Time Frame: Duration of recovery room stay (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
minutes | 30.3 (17.09) | 16.6 (8.38)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = 13.7, 95% CI 2-sided [0.63 to 26.77]

8. Secondary Outcome: First Pain Score in Recovery Room
Description: Pain was measured using an 11-point visual analogue scale (VAS). Range: 0-11 (0 = no pain; 11 = worst pain imaginable).
Time Frame: Duration of recovery room stay (average approximately 1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
score on a scale | 1.3 (2.41) | 1.3 (2.41)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 1, t-test, 2 sided; Mean Difference (Final Values) = 0, 95% CI 2-sided [-2.80 to 2.80]

9. Secondary Outcome: Discharge-ready Pain Score
Description: Pain was measured using an 11-point visual analogue scale (VAS). Range: 0-11 (0 = no pain; 11 = worst pain imaginable).
Time Frame: Day of discharge (up to 2 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
score on a scale | 1.1 (1.66) | 1.3 (2.26)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 0.82, t-test, 2 sided; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-2.38 to 1.98]

10. Secondary Outcome: Analgesic Consumption
Description: Analgesic consumption was measured in oral morphine milligram equivalents (MME)
Time Frame: Recovery room to 7th postoperative day
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
Number analyzed (Participants) | 10 | 10
MME | 0.5 (1.58) | 2 (4.83)
Statistical Analysis 1: Comparison: THRIVE vs Endotracheal Tube or Supraglottic Airway; Test type: Other; p = 0.37, t-test, 2 sided; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-5.29 to 2.29]

ADVERSE EVENTS:
Time Frame: Up to 1 week
Arm/Group | THRIVE | Endotracheal Tube or Supraglottic Airway
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT03086408/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT03086408/SAP_001.pdf